CLINICAL TRIAL: NCT00376987
Title: Do Dietary Supplements of Zinc Reduce Serum Cadmium Levels in Smokers?
Brief Title: Zinc Supplements in Lowering Cadmium Levels in Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000495325; CCCWFU-98903; CCCWFU-BG03-538
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-09

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: renal cell carcinoma; bladder cancer; cervical cancer; esophageal cancer; gastric cancer; adult acute myeloid leukemia; pancreatic cancer; hypopharyngeal cancer; lip and oral cavity cancer; laryngeal cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; non-small cell lung cancer; small cell lung cancer; adult primary liver cancer; tongue cancer; tobacco use disorder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Renal Cell; Leukemia, Myeloid, Acute; Hypopharyngeal Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular; Tongue Neoplasms | interventions — Zinc Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: zinc oxide — Oral daily dietary supplement containing 80 mg Zinc oxide

SUMMARY:
RATIONALE: Zinc supplements may lower cadmium levels in smokers and may help prevent DNA damage.

PURPOSE: This clinical trial is studying how well zinc supplements work in lowering cadmium levels in smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether zinc supplements reduce cadmium levels in smokers.
* Measure serum levels of cotinine (a biomarker of smoking), zinc (a marker of compliance), and cadmium (the dependent variable) at 3 pre-supplementation visits and at 6 supplementation visits.
* Determine whether serum cadmium levels (adjusted for serum levels of cotinine) decrease during supplementation with VisiVite Smoker's Formula.
* Determine if increased cadmium levels in the blood of cigarette smokers can be correlated with decreased mismatch repair.
* Determine if administration of zinc-containing supplements reverses cadmium-induced inhibition of mismatch repair.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive oral zinc supplements once daily for 12 weeks in the absence of unacceptable toxicity.

Blood, serum, and urine are collected once weekly for 3 weeks before beginning treatment and in weeks 5, 6, 9, 12, 15, and 17 for biomarker/laboratory analysis. Samples are examined for cadmium, zinc, and cotinine levels by atomic absorption spectrophotometry, expression of mismatch repair proteins (MSH2, MSH6, MSH3, MLH1, and PMS2), levels of messenger RNA by reverse transcriptase-polymerase chain reaction, and microsatellite instability by gel electrophoresis.

After completion of study therapy, patients are followed for 5 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently smoking ≥ 1 pack (20 cigarettes) per day
* Baseline cadmium level ≥ 0.5 μg/L

PATIENT CHARACTERISTICS:

* Negative pregnancy test
* Fertile patients must use effective contraception
* No known gastrointestinal upset due to zinc vitamins or lozenges

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior and no other concurrent vitamins and zinc supplements

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-12; Primary Completion 2006-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reduction of cadmium levels | 17 weeks
Serum levels of cotinine, zinc, and cadmium at 3 pre-supplementation visits and at 6 supplementation visits | 17 weeks
Correlation of increased cadmium levels with decreased mismatch repair | 17 weeks
Reversal of cadmium-induced inhibition of mismatch repair | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary G. Schwartz, MD, PhD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States